CLINICAL TRIAL: NCT06021080
Title: Effects of Different Continuous Renal Replacement Therapy Patterns on Ionized Calcium in Patients With Citrate Anticoagulants Using Calcium-containing Replacement Solutions
Status: Recruiting | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Han Chen, Deputy chief physician, Fujian Provincial Hospital
Other Study IDs: HChen
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-03

CONDITIONS: Renal Injury; Regional Citrate Anticoagulation; Continuous Renal Replacement Therapy
Keywords: Renal Injury; Regional citrate anticoagulation; Continuous renal replacement therapy
MeSH Terms: interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CVVHD: Continuous Veno-Venous Hemosdialysis
  Interventions: Procedure: CVVHD
- CVVH: Continuous Veno-Venous Hemofiltration
  Interventions: Procedure: CVVH

INTERVENTIONS:
Procedure: CVVH — CVVH therapy
  Groups: CVVH
Procedure: CVVHD — CVVHD therapy
  Groups: CVVHD

SUMMARY:
It is unclear whether different modes of continuous renal replacement therapy (CRRT) impact post-filter ionized calcium concentrations during regional citrate anticoagulation (RCA) when using calcium-containing replacement fluid.

This prospective, single-center, observational cohort study will screen all patients receiving CRRT for eligibility. General clinical information will be collected before commencing CRRT treatment. Patients will be randomly assigned to either the veno-venous hemofiltration (CVVH) or continuous veno-venous hemodialysis (CVVHD) group and switch to the alternative mode in the subsequent treatment session. Pre-filter and post-filter ionized calcium, systemic total and ionized calcium, and effluent total and ionized calcium will be measured 2 hours after the initiation of CRRT. Electrolyte levels, arterial blood gases, hourly citrate dose, and total citrate dose will be recorded every 6 hours until the end of CRRT. The primary outcome is the difference in ionized calcium concentrations at each site over time between the two modes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Receiving citrate anticoagulation;
3. Obtain Informed consent from patients or next of kin.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Allergic to citrate anticoagulants;
3. Severe liver dysfunction (total bilirubin levels exceeding two times the normal range);
4. Hypoxemia (PaO2 < 60 mmHg);
5. Inadequate tissue perfusion (blood pressure < 90/60 mmHg despite high doses of vasoactive agents);
6. Hyperlactatemia (lactate> 4 mmol/L);
7. Hypernatremia;
8. Estimated length of hospital stay < 48h;
9. Participated in other studies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU who need RCA-CRRT will be screened for study eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Post-filter iCa | 2 hours after the initiation of CRRT
  The post-filter ionized calcium concentration
Serum iCa | 2 hours after the initiation of CRRT
  Serum ionized calcium concentration
Serum Ca2+ | 2 hours after the initiation of CRRT
  Serum total calcium concentration
Effluent Ca2+ | 2 hours after the initiation of CRRT
  Effluent total calcium concentration

SECONDARY OUTCOMES:
Incidence of new-onset metabolic complications | 48 hours after the initiation of CRRT
  Including hypercalcemia, hypocalcemia, metabolic acidosis, metabolic alkalosis, citrate accumulation, hypernatremia, and hyponatremia

CONTACTS AND LOCATIONS:
Overall Officials: Han Chen, Ph.D., M.D., Principal Investigator — Fujian Provincial Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No